CLINICAL TRIAL: NCT02862340
Title: Study of the Involvement of 15q11 - q13 Chromosome Region and CYFIP1 Gene in Autism. Attempt a Genotype-phenotype Correlation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 07-PP-01
Record Dates: First submitted 2016-07-21; First posted 2016-08-11 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-08

CONDITIONS: Autistic Disorder
MeSH Terms: conditions — Autistic Disorder | interventions — Genetic Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Autistic disorder (Other): Children over 4 years with an autistic disorder of unknown etiology with the techniques currently available and accessible in routine diagnostics.
  Interventions: Genetic: Genetic test

INTERVENTIONS:
Genetic: Genetic test

SUMMARY:
Autism, ranked among the '' pervasive developmental disorders' (ASD), is characterized by disturbances in the areas of reciprocal social interaction, communication and behavior, interests and activities restricted, repetitive. Various studies indicate that autistic disorder is subjected to a genetic predisposition, most likely polygenic and heterogeneous. However, no major gene responsible for this disorder has yet been identified. Given the link between the Fragile X syndrome (the most common form of mental retardation (MR) hereditary) and autistic behavior, it seems interesting to look, also, a possible link to the molecular level. Among the proteins interacting with FMRP (absent protein in fragile X patients), the investigators were interested to CYFIP1, protein encoded by the gene CYFIP1 appears to be a good candidate gene involved in the RM and autism by its chromosomal position and function. As FMR1, CYFIP1 is expressed in the brain cortex, hippocampus and Purkinje cells of the cerebellum. This protein co-localizes and interacts with Rac and FMRP, which are both involved in neurogenesis and cognitive development. In humans, the gene encoding CYFIP1 is located in the 15q11-q13. Now, the only autosomal abnormalities most frequently observed in autism are those involving the proximal 15q region, including duplications or 15q11-q13 triplications interstitial, of maternal origin.

These data suggest that an / or more autism genes responsible are probably present in the 15q11-q13 chromosomal region, although no gene has yet been identified. Thus, the study of the role of CYFIP1 gene in patients with autism spectrum disorders would most likely contributory.

The investigators wish to study the involvement of the 15q11-q13 chromosomal region and CYFIP1 gene in autistic disorder in a hundred patients from the Autism Resource Centre (ARC) Nice PACA antenna, over a two year period.

The diagnosis and assessment report of children likely to be included in this study will be conducted at ARC Nice. Balance sheets are made according to the recommendations of the High Authority of Health for diagnosis of infantile autism and PDD. These children are then sent to the Genetic Consultation Nice Hospital where an analysis of the background and a specific morphological examination will be realized..

ELIGIBILITY:
Inclusion Criteria:

* Subject unadopted 4 to 18 years
* Subject completing the autism spectrum disorder criteria development by diagnostic grid ICD10 recognized by the international community child psychiatry. The ADI-R test is always associated.
* Subject has at least one of the following abnormalities:

Mental retardation, Anomaly morphological examination (abnormal weight and height growth and / or head circumference, abnormal ends, dysmorphic ...) Malformation (s) visceral (s) Behavioural disorders other than autistic disorder (aggression, sleep disorders ...) Abnormal neurological examination and brain imaging, Family history of autism and / or mental retardation.

- Parents of the subject and topics affiliated to a social security scheme

Exclusion Criteria:

* Etiologie de la pathologie autistique connue (Syndrome de Rett, Xfra…)
* Absence de consentement éclairé des patients et des représentants de l'autorité parentale
* Parents sous tutelle ou curatelle

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2008-01; Primary Completion 2008-01 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
presence or absence of abnormality in 15q11q13 gene | At the inclusion
  Testing a candidate gene in a chromosomal region known to be involved in autism

SECONDARY OUTCOMES:
phenotype | At the inclusion
  Syndromic or specific behavioral phenotypes corresponding to the identified molecular abnormalities

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nice, Nice, France

IPD SHARING:
Plan to Share IPD: No